CLINICAL TRIAL: NCT00533442
Title: Tacrolimus and Mycophenolate Mofetil vs Tacrolimus and Sirolimus in SPK, Pancreas After Kidney or Pancreas Transplant Alone
Brief Title: Rapamycin Versus Mycophenolate Mofetil in Kidney-Pancreas Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, George W. Burke, Professor of Surgery, University of Miami
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20000176
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes
Keywords: Rapamycin; Mycophenolate Mofetil (MMF); Kidney-Pancreas Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus; Mycophenolic Acid; Tacrolimus; Steroids; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus plus MMF plus Steroids (Active Comparator): Patients randomized to this arm were scheduled to receive maintenance therapy consisting of Tacrolimus, Mycophenolate Mofetil (MMF), and Steroids. Patients in both treatment arms received dual induction therapy consisting of Rabbit Anti-thymocyte Globulin (Thymoglobulin) plus Daclizumab.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Steroids
- Tacrolimus plus Rapamycin plus Steroids (Experimental): Patients randomized to this arm were scheduled to receive maintenance therapy consisting of Tacrolimus, Rapamycin (Sirolimus), and Steroids. Patients in both treatment arms received dual induction therapy consisting of Rabbit Anti-thymocyte Globulin (Thymoglobulin) plus Daclizumab.
  Interventions: Drug: Rapamycin; Drug: Tacrolimus; Drug: Steroids

INTERVENTIONS:
Drug: Rapamycin — Rapamycin was initiated on day 1 postoperatively, 4mg/day;levels were maintained 5-8ng/ml. Those patients randomized to receive mycophenolate mofetil were given 1gm twice/day starting on the first post-operative day.
  Other Names: Rapamune® (sirolimus)
  Arms: Tacrolimus plus Rapamycin plus Steroids
Drug: Mycophenolate Mofetil — MMF 1 gm BID beginning 1st day postoperative day
  Other Names: Cellcept; MMF
  Arms: Tacrolimus plus MMF plus Steroids
Drug: Tacrolimus — Part of standard maintenance.
  Other Names: TAC
Drug: Steroids — Part of standard maintenance
  Other Names: Corticosteroids

SUMMARY:
This study was designed to determine which maintenance immunosuppressive agent, rapamycin or mycophenalate mofetil, resulted in better outcome in patients with type 1 diabetes and renal failure, who presented for a kidney-pancreas transplant.

DETAILED DESCRIPTION:
This is a randomized, prospective single center study evaluating the two maintenance drugs above.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 1 diabetes and end stage renal disease.
* Women of childbearing potential must have had a negative pregnancy test (serum or urine).
* Patient agrees to participate in the study and sign an informed consent.
* Patient has no known contraindication to the administration of rapamycin or mycophenolate mofetil.
* Patient has no history of hypersensitivity to rapamycin or mycophenolate mofetil.

Exclusion Criteria:

* Patient has history of a malignancy within two years, with the exception of adequately treated localized squamous or basal cell carcinoma of the skin without evidence of recurrence.
* Patient is currently abusing drugs or alcohol.
* Patient is known or suspected to have an active infection or be seropositive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) or human immunodeficiency virus (HIV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2000-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W Burke, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Result] Burke GW 3rd, Ciancio G, Figueiro J, Olson L, Gomez C, Rosen A, Suzart K, Miller J. Steroid-resistant acute rejection following SPK: importance of maintaining therapeutic dosing in a triple-drug regimen. Transplant Proc. 2002 Aug;34(5):1918-9. doi: 10.1016/s0041-1345(02)03122-6. No abstract available. PMID 12176628
- [Result] Burke G 3rd, Ciancio G, Figueiro J, Olson L, Gomez C, Rosen A, Suzart K, Miller J. Can acute rejection be prevented in SPK transplantation? Transplant Proc. 2002 Aug;34(5):1913-4. doi: 10.1016/s0041-1345(02)03149-4. No abstract available. PMID 12176626
- [Result] Burke GW 3rd, Ciancio G, Figueiro J, Buigas R, Olson L, Roth D, Kupin W, Miller J. Hypercoagulable state associated with kidney-pancreas transplantation. Thromboelastogram-directed anti-coagulation and implications for future therapy. Clin Transplant. 2004 Aug;18(4):423-8. doi: 10.1111/j.1399-0012.2004.00183.x. PMID 15233820
- [Result] Ciancio G, Sageshima J, Chen L, Gaynor JJ, Hanson L, Tueros L, Montenora-Velarde E, Gomez C, Kupin W, Guerra G, Mattiazzi A, Fornoni A, Pugliese A, Roth D, Wolf M, Burke GW 3rd. Advantage of rapamycin over mycophenolate mofetil when used with tacrolimus for simultaneous pancreas kidney transplants: randomized, single-center trial at 10 years. Am J Transplant. 2012 Dec;12(12):3363-76. doi: 10.1111/j.1600-6143.2012.04235.x. Epub 2012 Sep 4. PMID 22946986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 1, 2000 through December 15, 2009, 170 consecutive patients with type 1 diabetes and ESRD were randomized to receive either Rapamycin (N=84) or MMF (N=86) immediately prior to transplant. Post-transplant clinical follow-up of patients continued through January 15, 2011.
Pre-assignment Details: A randomized block design was implemented for the randomization scheme using Proc Plan in SAS. Patients were randomly assigned (allocation ratio of 1:1) to the two treatment arms in blocks of 4 and 6 patients (block sizes were also chosen randomly), ensuring a balance of patients across treatment arms after each block of patients was randomized.
Groups:
- Tacrolimus Plus MMF Plus Steroids: This group of kidney-pancreas recipients was randomized to receive mycophenolate mofetil and tacrolimus after transplantation.
  Tacrolimus and mycophenolate mofetil: MMF 1 gm BID beginning 1st day postoperative day
- Tacrolimus Plus Rapamycin Plus Steroids: Patients randomized to this arm received Sirolimus, after kidney-pancreas transplantation.
  Rapamycin: Rapamycin was initiated on day 1 postoperatively, 4mg/day;levels were maintained 5-8ng/ml. Those patients randomized to receive mycophenolate mofetil were given 1gm twice/day starting on the first post-operative day.
  Rapamune and Tacrolimus: Sirolimus 2 mg/day beginning 1st postoperative day (trough target levels:
  10-15ng/ml)
  Mycophenolate Mofetil: Patients randomized to receive mycophenolate mofetil were given 1gm twice/day starting on the first post-operative day.
Period: Allocation and Intent to Treat Analysis
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids
Started | 86 | 84
Completed | 86 | 84
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids
Started | 86 (Ongoing Follow-up at 13-123 months (N=77); Lost to Follow-up (N=9, at 5-100 months).) | 84 (Ongoing Follow-up at 17-124 months (N=74); Lost to Follow-up (N=10, at 5-67 months).)
Completed | 77 | 74
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids | Total
Number analyzed (Participants) | 86 | 84 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (9.3) | 41.5 (8.2) | 42.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 55 | 50 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55 | 47 | 102
  Hispanic | 19 | 31 | 50
  African-American | 11 | 6 | 17
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-Specific Survival Comparisons
Description: Freedom from biopsy-proven acute rejection of the kidney allograft; Freedom from biopsy-proven acute rejection of the pancreas allograft; Death-censored kidney graft survival; Death-censored pancreas graft survival; Death-uncensored graft (kidney and pancreas) survival; and Patient survival.
Time Frame: over 1-10 years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids
Number analyzed (Participants) | 86 | 84
Participants
  Biopsy-Proven Acute Rejection of the Kidney | 22 | 8
  Biopsy-Proven Acute Rejection of the Pancreas | 9 | 1
  Death-Censored Kidney Graft Failure | 18 | 10
  Death-Censored Pancreas Graft Failure | 7 | 2
  Death-Uncensored Graft (Kidney&Pancreas) Survival | 26 | 25
  Patient Death | 16 | 15
Statistical Analysis 1: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Biopsy-Proven Acute Rejection of the Kidney (logrank test); Test type: Superiority; p = 0.01, Log Rank
Statistical Analysis 2: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Biopsy-Proven Acute Rejection of the Pancreas (logrank test); Test type: Superiority; p = 0.01, Log Rank
Statistical Analysis 3: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Death-Censored Kidney Graft Failure (logrank test); Test type: Superiority; p = 0.16, Log Rank
Statistical Analysis 4: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Death-Censored Pancreas Graft Failure (logrank test); Test type: Superiority; p = 0.12, Log Rank
Statistical Analysis 5: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Death-Uncensored (Kidney & Pancreas) Graft Survival (logrank test); Test type: Superiority; p = 0.96, Log Rank
Statistical Analysis 6: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Test type: Superiority; p > 0.99, Log Rank — Patient Death (logrank test)

2. Secondary Outcome: Overall Kidney Transplant Function at 12, 36, and 60 Months Post-transplant.
Description: Comparisons of renal function (eGFR, measured in mL/min/1.73 m^2) at 12, 36, and 60 months post-transplant.
Time Frame: at 1-5 years post-transplant
Population: Number analyzed here includes all patients alive with a functioning graft that had an available measurement taken at that time
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus Plus Rapamycin Plus Steroids | Tacrolimus Plus MMF Plus Steroids
Number analyzed (Participants) | 84 | 86
mL/min/1.73m^2
  Mean eGFR at 12 months: number analyzed (Participants) | 75 | 78
  Mean eGFR at 12 months | 71.2 (2.4) | 67.2 (2.0)
  Mean eGFR at 36 months: number analyzed (Participants) | 60 | 62
  Mean eGFR at 36 months | 63.0 (3.1) | 61.5 (2.6)
  Mean eGFR at 60 months: number analyzed (Participants) | 38 | 43
  Mean eGFR at 60 months | 56.5 (4.1) | 61.9 (3.8)
Statistical Analysis 1: Comparison: Tacrolimus Plus Rapamycin Plus Steroids vs Tacrolimus Plus MMF Plus Steroids; Comparison of Mean eGFR at 12 Months Post-Transplant (t-test); Test type: Superiority; p = 0.21, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus Plus Rapamycin Plus Steroids vs Tacrolimus Plus MMF Plus Steroids; Comparison of Mean eGFR at 36 Months Post-Transplant (t-test); Test type: Superiority; p = 0.71, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus Plus Rapamycin Plus Steroids vs Tacrolimus Plus MMF Plus Steroids; Comparison of Mean eGFR at 60 Months Post-Transplant (t-test); Test type: Superiority; p = 0.33, t-test, 2 sided

3. Secondary Outcome: Overall Pancreas Transplant Function at 12, 36, and 60 Months Post-transplant.
Description: Comparisons of pancreas function (C-peptide in ng/mL) at 12, 36, and 60 months post-transplant.
Time Frame: at 1-5 years post-transplant
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids
Number analyzed (Participants) | 86 | 84
ng/mL
  Mean Log {C-peptide at 12 months}: number analyzed (Participants) | 53 | 61
  Mean Log {C-peptide at 12 months} | 1.15 (0.08) | 1.08 (0.07)
  Mean Log {C-peptide at 36 months}: number analyzed (Participants) | 45 | 43
  Mean Log {C-peptide at 36 months} | 0.990 (0.08) | 0.986 (0.08)
  Mean Log {C-peptide at 60 months}: number analyzed (Participants) | 33 | 34
  Mean Log {C-peptide at 60 months} | 1.17 (0.10) | 1.22 (0.10)
Statistical Analysis 1: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Comparison of Mean Log {C-Peptide Level} at 12 Months Post-Transplant (t-test); Test type: Superiority; p = .47, t-test, 2 sided
Statistical Analysis 2: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Comparison of Mean Log {C-Peptide Level} at 36 Months Post-Transplant (t-test); Test type: Superiority; p = 0.97, t-test, 2 sided
Statistical Analysis 3: Comparison: Tacrolimus Plus MMF Plus Steroids vs Tacrolimus Plus Rapamycin Plus Steroids; Comparison of Mean Log {C-Peptide Level} at 60 Months Post-Transplant (t-test); Test type: Superiority; p = 0.75, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: during the first year post-transplant
Description: Serious Adverse Events were defined as: 1) the occurrence of any infection that required hospitalization, and 2) a major cardiovascular event.
Arm/Group | Tacrolimus Plus MMF Plus Steroids | Tacrolimus Plus Rapamycin Plus Steroids
All-Cause Mortality (participants affected / at risk) | 16/86 | 15/84
Serious Adverse Events (participants affected / at risk) | 40/86 | 38/84
Other Adverse Events (participants affected / at risk) | 3/86 | 5/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus Plus MMF Plus Steroids (N=86) | Tacrolimus Plus Rapamycin Plus Steroids (N=84)
Infection (Infections and infestations) | 31 (31) | 32 (32)
Major Cardiovascular Event (Vascular disorders) | 15 (15) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus Plus MMF Plus Steroids (N=86) | Tacrolimus Plus Rapamycin Plus Steroids (N=84)
New Onset Diabetes Mellitus Type 2 after Transplant (NODAT) (Endocrine disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No